CLINICAL TRIAL: NCT05267847
Title: The Success Rate of Cryotherapy Application in Primary Molars With Signs of Irreversible
Brief Title: The Success Rate of Cryotherapy Application in Primary Molars With Signs of Irreversible Pulpitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Assistant Professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 133
Record Dates: First submitted 2022-02-22; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy during inferior alveolar nerve block (Experimental)
  Interventions: Other: Cryotherapy
- Inferior alveolar nerve block (Active Comparator)
  Interventions: Other: Traditional local anesthesia

INTERVENTIONS:
Other: Cryotherapy — local anesthetic injection with articaine 4% 1:100,000 epinephrine then an application ice packs
  Arms: Cryotherapy during inferior alveolar nerve block
Other: Traditional local anesthesia — local anesthetic injection with articaine 4% 1:100,000 epinephrine
  Arms: Inferior alveolar nerve block

SUMMARY:
The study is designed as a randomized controlled trial with two parallel groups. Children aged 5-9 years with primary molars from suffered symptomatic signs of irreversible pulpitis will be randomly assigned into two groups. The first group (experimental group) will be injected with 4% articaine 1:100.000 epinephrine (inferior alveolar nerve block). For the second group, the mandibular second primary molars will be anesthetized using 4% articaine 1:100.000 epinephrine using inferior alveolar nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children are classified as I or II according to ASA
* Presence of at least one mandibular primary molar with symptomatic signs of irreversible pulpitis
* Presence of at least two-thirds of the root length in periapical radiograph

Exclusion Criteria:

* Unrestorable crowns
* Children with systemic, severe behavior or emotional problems
* Presence of gingival redness, swellings, fistulous of sinus tract
* Radiographic evidence of internal root resorption, pulp stones or calcifications, and/or bone radiolucency

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2022-02-22 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | up to 24 hours
  Wong Backer pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Ahmed, Al Minyā, Egypt

REFERENCES:
- [Derived] Elheeny AAH, Sermani DI, Saliab EA, Turky M. Cryotherapy and pain intensity during endodontic treatment of mandibular first permanent molars with symptomatic irreversible pulpitis: A randomized controlled trial. Clin Oral Investig. 2023 Aug;27(8):4585-4593. doi: 10.1007/s00784-023-05084-1. Epub 2023 Jun 3. PMID 37268843